CLINICAL TRIAL: NCT01366118
Title: Prospective Pilot Study of Therapeutic Targets (TT) Tailored Chemotherapy (Ch) and Intensity Modulated Radiotherapy (IMRT) as Neoadjuvant Treatment in Patients With Rectal Carcinoma
Brief Title: Study of Therapeutic Targets Tailored Ch and IMRT as Neoadjuvant Treatment in Rectal Carcinoma Patients
Acronym: TT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Hospital de Madrid (Other)
Responsible Party: Fundación Hospital de Madrid, Centro Integral Oncológico Clara Campal
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62 202-878
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2009-10

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer, Chemoradiotherapy, target therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TT tailored Ch plus IMRT (Experimental)
  Interventions: Drug: Therapeutic target tailored chemotherapy

INTERVENTIONS:
Drug: Therapeutic target tailored chemotherapy — All pts were treated with Capecitabine (Cap) 625-825 mg/m2/12h M-F.
  Ch combination schema was customized based on:
  Top- 1 +: Irinotecan (I) 50mg/m2 / in weekly. Top-1 - and ERCC-1 - : Oxaliplatin (O) 50gm/m2/ weekly. Top- 1 - and ERCC-1 + : Neither I nor O. K-Ras or b-Raf mutated (m) : Bevacizumab (B) 5mg/kg every two weeks. K-Ras and B-Raf native (n): Cetuximab (C) 400/250mg/m2 weekly or B (investigator option). Figure 1.
  When Cap was in combination with O or I the 625mg/m2 dose was chosen. When Cap was the only chemotherapy agent in combination with B or C the 825mg/m2 dose was chosen
  Other Names: Therapeutic targets; Oxaliplatin; CPT-11; 5-FU

SUMMARY:
The parameter that best correlates with 5 years disease-free survival (DFS ) in patients (pts) with localized rectal cancer (RC) is the pathological TNM staging (ypTNM) after chemo-radiotherapy (Ch-RT). DFS is 97% in pts with ypT0N0M0 = ypCR and 42% in pts with ypN +. Standard 5-FU Ch-RT achieves 15% of ypCR. The use of IMRT achieves a high proportion of ypCR . This study aimed to demonstrate in a prospective manner the feasibility of personalizing Ch regimen base in TT in combination with IMRT in patients with RC. Secondary objectives included the number of ypCR and safety.

DETAILED DESCRIPTION:
The parameter that best correlates with DFS in patients (pts) with localized rectal cancer (RC) is the pathological TNM staging (ypTNM) after chemo-radiotherapy (Ch-RT).Tumor regression grading (TRG) after Ch-RT has been correlated with DFS , 86% for TRG 4, 75% for grouped TRG 2 + 3, and 63% for grouped TRG 0 + 1 but this is not as good as ypTNM to predict pts outcome.

Standard 5-FU or capecitabine Ch-RT achieves 15% of ypCR with diarrhea and proctitis as the main grade 3 toxicities in the range of 10-15% . With the combination of oxaliplatin and capecitabine pCR rates are the same but the toxicity is the range of 25%. IMRT studies reported 30% ypCR but with 30-40% grade 3 toxicities Last years strategies have explored ways to integrate additional chemotherapeutic agents as capecitabine , oxaliplatin, irinotecan, bevacizumab and cetuximab in Ch-RT regimens and to find biomarkers of their effectiveness , but always in a retrospective way.

Our hypothesis is that with the actual knowledge and technology, a prospective tailored chemotherapy selection in combination with IMRT is feasible and could improve the outcome of patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of rectal adenocarcinoma.
* Clinical stage II or III.
* Feasible patient for neoadjuvant Ch-RT.
* Availability of tumor tissue or possibility of a tumor biopsy to define therapeutic targets.
* Informed written consent was obtained from all patients

Exclusion Criteria:

* Contraindication to the administration of any of the drugs used in the study capecitabine, irinotecan, oxaliplatin, cetuximab or bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
ypTN | Up to 1 month
  pathology TN after neoadjuvant treatment and surgery

SECONDARY OUTCOMES:
Feasibility | Up to 3 months
  Days needed to full set of TT analys. Days from signed informed consent to first day of Ch-RT treatment Number of patinets who complet the Ch-RT treatment and go to surgery as planned.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD.PhD, Principal Investigator — Centro Integral Oncológico Clara Campal
Locations (1):
- Centro Integral Oncológico Clara Campal, Madrid, Madrid, Spain